CLINICAL TRIAL: NCT06334133
Title: Cadisegliatin as Adjunctive Therapy in Type 1 Diabetes: A 26-Week Double-Blind, Randomized, Placebo-Controlled Phase 3 Study
Brief Title: Cadisegliatin as Adjunctive Therapy to Insulin in Participants With Type 1 Diabetes
Acronym: CATT1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: vTv Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TTP399-302
Record Dates: First submitted 2024-03-13; First posted 2024-03-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — TTP399; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cadisegliatin: 26 Week Double Blind Treatment Period - 800 mg QD (Experimental): The main study uses a randomized, double-blind, placebo-controlled design with parallel assignment among 3 treatment arms. The trial begins with a screening period of up to 14 days, followed by a 28-day device training and insulin adjustment period leading into a 28-day baseline period before entering the 26-week treatment period. Insulin is adjunctive therapy.
  Interventions: Drug: Cadisegliatin 800 mg QD
- Cadisegliatin: 26 Week Double Blind Treatment Period - 800 mg BID (Experimental): The main study uses a randomized, double-blind, placebo-controlled design with parallel assignment among 3 treatment arms. The trial begins with a screening period of up to 14 days, followed by a 28-day device training and insulin adjustment period leading into a 28-day baseline period before entering the 26-week treatment period. Insulin is adjunctive therapy.
  Interventions: Drug: Cadisegliatin 800 mg BID
- Placebo: 26 Week Double Blind Treatment Period (Placebo Comparator): The main study uses a randomized, double-blind, placebo-controlled design with parallel assignment among 3 treatment arms. The trial begins with a screening period of up to 14 days, followed by a 28-day device training and insulin adjustment period leading into a 28-day baseline period before entering the 26-week treatment period. Insulin is adjunctive therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cadisegliatin 800 mg QD — Cadisegliatin is an orally bioavailable small-molecule glucokinase activator; adjunctive therapy to insulin.
  Other Names: TTP399
  Arms: Cadisegliatin: 26 Week Double Blind Treatment Period - 800 mg QD
Drug: Cadisegliatin 800 mg BID — Cadisegliatin is an orally bioavailable small-molecule glucokinase activator; adjunctive therapy to insulin.
  Other Names: TTP399
  Arms: Cadisegliatin: 26 Week Double Blind Treatment Period - 800 mg BID
Drug: Placebo — Placebo (insulin alone)
  Arms: Placebo: 26 Week Double Blind Treatment Period

SUMMARY:
This is a Phase 3 trial of cadisegliatin as adjunctive therapy to insulin in participants with Type 1 Diabetes Mellitus.

DETAILED DESCRIPTION:
Study TTP399-302 is a 26-week, Phase 3 trial designed to measure the relative efficacy of adjunctive treatment with cadisegliatin to reduce the incidence of Level 2 or Level 3 hypoglycemia in participants with Type 1 Diabetes Mellitus compared to placebo (insulin alone) over 26 weeks of continuous therapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥18 years
* Diagnosed T1DM with a minimum of 3 years since diagnosis
* Has had at least 1 hypoglycemic event of Level 2 (glucose level <54 mg/dL or <3 mmol/L, [CGM or SMBG confirmed]) or Level 3 (defined as a severe hypoglycemia with altered mental state and/or physical status requiring assistance) in the last 2 months prior to Screening
* HbA1c value of <9.5% at Screening
* Is currently on CSII (closed-loop systems are prohibited) or is on MDI for at least 6 months prior to the Screening Visit and is willing to stay on same type of insulin treatment and the current mode of insulin administration (CSII or MDI injection treatments) for the duration of the study
* Must have been on a CGM device for at least 3 months prior to Screening

Exclusion Criteria:

* Has T2DM, monogenic diabetes, maturity-onset diabetes of the young, other unusual or rare forms of diabetes mellitus, or diabetes resulting from a secondary disease
* Has been hospitalized for DKA within 3 months prior to Screening
* Has uncontrolled hypothyroidism or hyperthyroidism
* History of eating disorder within the last 2 years such as anorexia, bulimia, diabulimia or neglecting to give insulin to manipulate weight
* Has an active or untreated malignancy, or has been in remission from malignancy for ≤5 years except well-treated basal cell or squamous cell skin cancer or cervical cancer in situ
* Has used any of the following medications within the specified time periods - any non-insulin anti-diabetic therapies, e.g., sodium glucose cotransporter-2 (SGLT-2) inhibitors, glucagon-like peptide-1 (GLP-1) receptor agonists, metformin, sulfonylureas, dipeptidyl peptidase-4 (DPP-4) inhibitors, or pramlintide, alpha-glucosidase inhibitors, or glucose-dependent insulinotropic polypeptide agonists) or weight loss medications within 30 days prior to the Screening
* Has used a hybrid closed-loop system (e.g., Medtronic 670G, Omnipod 5, or Tandem X2 with control IQ) or Do-It-Yourself looping within the last 30 days prior to the Screening Visit, and agrees to not start hybrid closed-loop systems or Do-It-Yourself looping during the study.
* Has an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 utilizing the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at Screening
* Has uncontrolled hypertension prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in incidence of Level 2 or Level 3 hypoglycemia | 26 weeks
  Number of events of Level 2 or Level 3 hypoglycemia in participants on cadisegliatin vs placebo.

SECONDARY OUTCOMES:
To assess the change in HbA1c | 26 weeks
  Change from baseline in HbA1c in participants on cadisegliatin vs placebo.
To assess the effects of treatment on CGM-based metrics for glycemic control | 26 weeks
  Change from baseline for time in, above or below target range of participants on cadisegliatin vs placebo
To assess the effects of treatment on the incidence of diabetic ketoacidosis | 26 weeks
  Number of events of diabetic ketoacidosis participants on cadisegliatin vs placebo
To assess the effects of treatment on insulin dosing | 18 weeks
  Change from baseline in average daily total insulin on cadisegliatin vs placebo
To assess the effects of treatment on body weight | 26 weeks
  Change from baseline in mean body weight
To assess the incidence of treatment emergent adverse events | 26 weeks
  Number of treatment emergent adverse events with cadisegliatin vs placebo
To assess the incidence of treatment emergent adverse events leading to discontinuation | 26 weeks
  Number of treatment emergent adverse events leading to discontinuation with cadisegliatin vs placebo
To assess the incidence of adverse events of special interest | 26 weeks
  Number of adverse events of special interests with cadisegliatin vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Strack, MD, Study Director — vTv Therapeutics
Locations (45):
- United States (45):
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Advanced Metabolic Care & Research Institute, Inc. (AMCR), Escondido, California
  - MD Studies, Inc, Fountain Valley, California
  - AME Clinical Research, Huntington Beach, California
  - 310 Clinical Research, Inglewood, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Paradigm Clinical Research - Modesto, Modesto, California
  - Amicis Research Center, Northridge, California
  - Paradigm Clinical Research Centers LLC, San Diego, California
  - Acclaim Clinical Research, San Diego, California
  - Focus Clinical Research, West Hills, California
  - Denver Endocrinology Diabetes and Thyroid Center, Englewood, Colorado
  - BayCare Health Systems, Clearwater, Florida
  - ALL Medical Research, LLC, Cooper City, Florida
  - Excellence Medical and Research, Miami Gardens, Florida
  - Metabolic Research Institute, Inc, West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - East Coast Institute for Research, LLC, Canton, Georgia
  - Centricity Research - Columbus, Columbus, Georgia
  - The Jones Center Clinical Research, LLC, Macon, Georgia
  - Endocrine Research Solutions, Inc, Roswell, Georgia
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Johnson County Clin-Trials, LLC, Lenexa, Kansas
  - Profound Research LLC, Farmington Hills, Michigan
  - Excel Clinical Research, Las Vegas, Nevada
  - Palm Research Center, Las Vegas, Nevada
  - Vector Clinical Trials, Sparks, Nevada
  - Jacobi Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Javarra Inc., Charlotte, North Carolina
  - Physician's East PA, Greenville, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Diabetes & Endocrinology Associates of Stark County, Inc, Canton, Ohio
  - John Muir Physician Network Clinical Research Center, Concord, Ohio
  - Velocity Clinical Research - Medford, Medford, Oregon
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Texas Diabetes and Endocrinology, P.A, Austin, Texas
  - Velocity Clinical Research - Dallas, Dallas, Texas
  - Southern Endocrinology Associates PA, Mesquite, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Advanced Research Institute - Ogden, Ogden, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - University of Washington Diabetes Institute, Seattle, Washington

REFERENCES:
- See also: T1D Exchange prescreening website — https://t1dexchange.org/vtv-therapeutics-study/